CLINICAL TRIAL: NCT05685251
Title: Staying Healthy After Childbirth: My Hypertension Education and Reaching Target Program for Postpartum (STAC-MyHEARTp)
Brief Title: Staying Healthy After Childbirth: My Hypertension Education and Reaching Target Program for Postpartum
Acronym: STAC-MyHEARTp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Meriter Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2025-0768; Protocol Version 5/9/2024 (Other: UW Madison)
Record Dates: First submitted 2023-01-05; First posted 2023-01-17 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-04

CONDITIONS: Hypertension
Keywords: postpartum; chronic hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: A randomized, single-center study
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Coaching (Experimental)
  Interventions: Other: Health Coaching; Other: Home Blood Pressure Monitoring
- Standard of Care (No Intervention)

INTERVENTIONS:
Other: Health Coaching — Participants will receive a health coach telehealth/video visit or phone call every 2 weeks for 4 months, for a total of 8 calls. After these initial 8 calls, at approximately 6 months postpartum, the health coach will schedule maintenance calls 1 per month until approximately 12 months postpartum, for a total of 6 additional calls.
  Arms: Health Coaching
Other: Home Blood Pressure Monitoring — Participants will be provided an A&D UA-651 (BT) home blood pressure monitor with an appropriate cuff size, they will be asked to take their blood pressure at least three days a week, 2 measurements each time
  Arms: Health Coaching

SUMMARY:
A study of Staying Healthy After Childbirth (STAC) and My Hypertension Education And Reaching Target (MyHEART) for postpartum (p) patients to determine if health coaching can increase 12-month postpartum care attendance, hypertension control and hypertension self-management behavior compared to usual clinical care in patients with chronic hypertension or persistent pregnancy associated hypertension - postpartum. 140 participants will be enrolled and can expect to be on study for 12 months.

DETAILED DESCRIPTION:
To address the critical need for hypertension (HTN) control in young adults, the investigators developed the MyHEART (My Hypertension Education And Reaching Target) program, a multi-component patient-centered, theoretically-based intervention designed to increase self-management using evidence-based health behavior approaches to lower BP among young adults with uncontrolled HTN.

A nonrandomized, single-center pilot study of MyHEART was conducted, which established feasibility, satisfaction, and informed the design of this trial. A large, multi-site randomized-controlled trial to evaluate the effect of MyHEART (home blood pressure monitor distribution and heath coaching) on clinical outcomes, the change in systolic and diastolic blood pressure (primary) and HTN control (secondary) after 6 and 12 months, compared to usual clinical care was completed. Additionally, lifestyle changes and HTN self-management behavior were evaluated.

Incorporating components of the MyHEART intervention with routine clinical care can support HTN behavioral changes in young adults with uncontrolled HTN to support BP lowering in this population. The investigators are in a unique position to partner with the Perinatal Clinic and the current STAC program, to improve health outcomes for women with HTN during pregnancy through health coaching and BP surveillance through 12-months postpartum.

Specific Aims:

* Aim 1: To improve postpartum attendance for 12-month hypertension follow-up care among Staying Healthy After Childbirth patients who have chronic hypertension or persistent hypertension at 6-weeks postpartum.

  * Hypothesis: Postpartum follow up care will improve in the intervention compared to usual care.
* Aim 2: To improve blood pressure control at 12-months in postpartum patients with chronic hypertension or a hypertension disorder of pregnancy with persistent HTN at 6-weeks postpartum.

  * Hypothesis: Blood pressure control will improve in the intervention (health coaching) arm compared to the usual care arm, via chart review from the 12-month postpartum appointment, and on ambulatory blood pressure monitoring compared to usual care.
* Aim 3: To increase lifestyle modification behaviors and health outcomes relating to nutrition and physical activity and cardiovascular disease (CVD) prevention in postpartum patients with chronic hypertension or a hypertension disorder of pregnancy with persistent HTN at 6-weeks postpartum.

  * Hypothesis: Health outcomes including, weight, lipid profile, A1c and microalbumin creatine ratio will improve in the intervention compared to usual care arm, via study surveys and upon chart review from the 12-month postpartum appointment.

Aim 1-3: A total of 140 participants will be enrolled and randomly assigned to the intervention and usual care arms.

ELIGIBILITY:
Inclusion Criteria:

* Willing and capable of giving written informed consent
* Willing to comply with all study procedures and be available for the duration of the study
* Genetically female
* Patients who complete the 6-week program, had a hypertension disorder of pregnancy who have persistent hypertension (systolic blood pressure greater than 130 mmHg or diastolic blood pressure greater than 80 mmHg) and/or are still on antihypertensive medication and those with chronic hypertension (CHTN) will be eligible to participate.
* Medically homed at UW Health or UPH

Exclusion Criteria:

* Inability to participate in health coaching (i.e., no reliable phone contact or Wi-Fi
* History of medically determined Congestive Heart Failure
* Unable to provide informed consent (i.e., activated healthcare power of attorney)
* Unable or unwilling to travel to local clinic for research visits
* Currently residing in a skilled nursing facility
* Diagnosed with sickle cell anemia or cystic fibrosis
* Diagnosed with stroke, myocardial infarction, and/or coronary artery revascularization in the past 2 years
* Syncope while exercising or doing strenuous activity within past 12 months
* Currently prescribed warfarin, novel oral anticoagulant, or insulin
* Planned organ transplant or prior transplant in the past 5 years
* Chemotherapy or radiation therapy within 6 the past months
* Severely impaired hearing, vision, or speech, as determined by study staff responsible for enrollment
* Current participation or planning to participate in another clinical trial in the next 12 months that involves hypertension management/control
* Pregnant or planning to become pregnant in the next 12 months
* Planning to leave the geographic area in the next 12 months
* Health condition that will limit both increasing physical activity and changing diet
* Illegal drug use (other than marijuana) in the past 30 days
* Unable to read or communicate in English
* Currently on dialysis or seeing a Nephrologist
* Unaware or denies history of high blood pressure or hypertension
* Between-arm blood pressure difference >20 mmHg
* Inability to comply with or complete the protocol or other reasons at the discretion of the principal and site investigators
* Prisoners

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants Who Attend 12 month Postpartum Care Visit | up to 12 months

SECONDARY OUTCOMES:
Difference in Self-Reported and Electronic Medical Record (EMR) documented BP at 6 months postpartum | up to 6 months
Lipid Profile at 12 months postpartum | 12 months
Hemoglobin A1c at 12 months postpartum | 12 months
Microalbumin Creatine Ratio at 12 months postpartum | 12 months
Percentage of participants that achieve hypertension control at 12 months postpartum | 12 months
  Hypertension control will be defined using ambulatory blood pressures as the gold standard (less than 130/80 mmHg); otherwise a clinic blood pressure of less than 140/90 mmHg will be used.
Hypertension Control: Number of Participants who initiate, titrate, or cease BP medications | up to 12 months
Hypertension Control: Summary of Antihypertensive Type | up to 12 months
Dietary Changes: Change in Sodium intake (milligrams/day) as assessed by the Automated Self-Administered 24-hour Dietary Assessment | 6 and 12 months
  Change in hypertension self-management behavior at 6 and 12 months compared to usual care will in part be assessed by dietary changes documented on an automated self-administered 24 hour dietary assessment.
Change in physical activity as measured by the Godin Physical Activity Questionnaire | 6 and 12 months
  Change in hypertension self-management behavior at 6 and 12 months compared to usual care will in part be assessed by change in physical activity as measured by the Godin Physical Activity Questionnaire at 6 and 12 months. The Godin Physical Activity Questionnaire measures a person's strenuous, moderate, and light physical activity in a week. A score of less than 14 is interpreted as insufficiently active or sedentary, a score between 14 and 23 is interpreted to be moderately active, and a score of 24 and higher is interpreted to be active.
Change in Home Blood Pressure Monitoring Frequency | 6 and 12 months
  Change in hypertension self-management behavior at 6 and 12 months compared to usual care will in part be assessed by measuring the frequency of home blood pressure monitoring.
Change in Weight (kg) | 6 and 12 months
  Change in hypertension self-management behavior at 6 and 12 months compared to usual care will in part be assessed by documenting participant weight at 6 and 12 months.
Change in Body Mass Index (BMI) | 6 and 12 months
  Change in hypertension self-management behavior at 6 and 12 months compared to usual care will in part be assessed by documenting participant BMI at 6 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Kara K Hoppe, DO, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- UW Hospital and Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes